CLINICAL TRIAL: NCT01311128
Title: Determination of the Accuracy of a Non-Invasive Continuous Blood Pressure Device
Status: Terminated | Type: Observational
Why Stopped: PI left institution
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Other Study IDs: 6980
Record Dates: First submitted 2011-03-08; First posted 2011-03-09 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Critically Ill
Keywords: Blood pressure; Heart rate; Cardiac output; Critical care; Perioperative care
MeSH Terms: conditions — Critical Illness | interventions — Mutagenesis, Insertional; Hemodynamic Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Heart rate and blood pressure determination: All subjects have the same conditions (T-line, blood pressure cuff, and radial artery catheter), in order to compare them within-subjects.
  Interventions: Device: T-line hemodynamic monitoring device (placement and use)

INTERVENTIONS:
Device: T-line hemodynamic monitoring device (placement and use) — The T-line device will be placed over the contralateral (from the radial artery catheter) radial artery at the distal wrist. To attach the device, a single-use sterile sensor is placed over the radial artery and the device then gently clamped around the wrist to incorporate the sensor. After a ten-minute stabilization period, data will be recorded every ten minutes during the first two hours of surgery, or until the patient is placed on cardiopulmonary bypass. The T-line device will then be removed. This procedure will be repeated, for a second two-hour period, in the ICU postoperatively.
  Other Names: T-line; Tensymeter; Tensys Medical, Inc.; Hemodynamic monitoring

SUMMARY:
This protocol will test a new non-invasive device, the T-line, in continuously determining heart rate and blood pressure in operative and critically ill patients. The accuracy of the device will be compared to the standard radial artery catheter, as well as to the non-invasive blood pressure cuff. The T-line will also be compared to the right heart catheter determining cardiac output in at least 20 patients.

Hypothesis: the T-line device will determine blood pressure and heart rate as accurately as a standard radial arterial catheter and a blood pressure cuff in perioperative patients.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years old
* Operative patients expected to require intensive care recovery at OHSU
* Planned or existing intra- and postoperative radial artery catheterization as part of routine care
* Palpable contralateral (to catheter) radial artery pulse
* Planned intraoperative right heart catheter placement as part of routine clinical care, in at least 20 subjects of total

Exclusion Criteria:

* No palpable radial artery pulse
* Anatomical abnormalities (skin grafts, cysts, cellulitis) or injuries (scarring, cuts, burns, bruising) at the sensor site
* An intravenous line placed at the sensor application site or within the medial/lateral travel range of the sensor
* An AV shunt in the T-line arm
* Known sensitivity to pressure stimuli (dermatographism)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-02-16 (Actual); Primary Completion 2012-06-29 (Actual); Study Completion 2014-12-30 (Actual)

PRIMARY OUTCOMES:
Agreement between radial catheter, blood pressure cuff, and T-line in determining heart rate and blood pressure | Assessed 24 times over four hours

SECONDARY OUTCOMES:
Agreement between the T-line and right heart catheter in determining cardiac output | Assessed every 30 minutes over four hours

CONTACTS AND LOCATIONS:
Overall Officials: Charles Phillips, MD, Principal Investigator — 503-494-2465
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States